CLINICAL TRIAL: NCT06888882
Title: Dilated Perivascular Spaces in the Dentate Nucleus on MRI in Patients with Hypertensive Angiopathy or Cerebral Amyloid Angiopathy
Acronym: HA-DN-DPVS
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2025/DR-02
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hypertensive Arteriopathy; Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CAA: Patients with cerebral amyloid angiopathy
- HA: Patients with Hypertensive arteriopathy

SUMMARY:
Hypertensive arteriopathy (HA) and cerebral amyloid angiopathy (CAA) are the two most common forms of cerebral small vessel disease. On MRI, chronic small vessel disease-related abnormalities include white matter hyperintensities, dilated perivascular spaces (DPVS), lacunar infarction, and hemorrhagic features (e.g. cerebral microbleeds, CMB). In the cerebellum, deep CMB involving the dentate nucleus (DN) is associated with HA, whereas the presence of superficial cerebellar CMB are associated with CAA. DPVS are observed in both diseases, predominant in the subcortical white matter (especially in the centrum semiovale) in CAA whereas HA-related DPVS are predominant deep in the brain inside or nearby the basal ganglia.

To the best of our knowledge, DN-DPVS have never been studies systematically in small vessel disease. The researchers want to study DN-DPVS on T2-weighted 3T MRI in patients with HA or CAA and to compare both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient registered in the CHU de Nîmes (France) stroke database with lobar intracerebral hemorrhage [ICH], subarachnoid hemorrhage or cortical superficial siderosis for CAA or basal ganglion ICH for HA
* Patient managed at the CHU de Nîmes (France) between 01/1/2015 and 31/12/2024
* Patient with T2-weighted MRI performed with a 3T magnet

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lobar intracerebral hemorrhage [ICH], subarachnoid hemorrhage or cortical superficial siderosis for CAA or basal ganglion ICH for HA
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sex | baseline
  Comparaison of both populations (HA/CAA), H/F
Hypertension | baseline
  history of hypertension (Yes/No)
Age | baseline
  Age at time of T2-weighted imaging,
Time | baseline
  Time between initial MRI-based CAA/HA diagnosis and 3T T2-weighted imaging, axial or coronal views of T2 imaging,
MRI view | baseline
  T2 performed using coronal or axial imaging (axial / coronal
hypercholesterolemia | baseline
  history of hypercholesterolemia (Yes/No)
Hemorrhagic lesion | baseline
  Hemorrhagic lesion load on T2*-weighted imaging (ICH and CMB for both CAA and HA, and subarachnoid hemorrhage/cortical superficial siderosis for CAA)
Subcortical lobar DPVS | baseline
  Semi-quantitative score for evaluation of subcortical lobar DPVS (0 if DPVS are absent, 1 if 1 to 10 DPVS are visible, 2 for 11 to 20 DPVS, 3 for 21 to 40 DPVS, and 4 for >40 DPVS).
DPVS of basal ganglia | baseline
  Semi-quantitative score for evaluation of DPVS of basal ganglia (0 if DPVS are absent, 1 if 1 to 10 DPVS are visible, 2 for 11 to 20 DPVS, 3 for 21 to 40 DPVS, and 4 for >40 DPVS).
Diabete | baseline
  history of diabetes (Yes/No)
Smoking | Baseline
  current smoking (Yes / No)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, Occitanie, France